CLINICAL TRIAL: NCT03158896
Title: A Phase I Study To Evaluate the Safety of Umbilical Cord - Derived, Ex-Vivo Cultured and Expanded Wharton's Jelly Mesenchymal Stem Cells for the Treatment of De Novo High Risk Acute or Steroid Refractory Acute Graft Versus Host Disease
Brief Title: Evaluation of Umbilical Cord-Derived Wharton's Jelly Stem Cells for the Treatment of Acute Graft Versus Host Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2016-aGvHD-MSCTC-0010
Record Dates: First submitted 2017-05-16; First posted 2017-05-18 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Acute Graft Versus Host Disease
Keywords: mesenchymal stem cell; hematopoietic stem cell transplant; Allogeneic hematopoietic stem cell transplant; Autologous hematopoietic stem cell transplant; Wharton's jelly; umbilical cord blood; steroid refractory graft versus host disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MSCTC-0010 Dose Escalation (Experimental): Cohort 1: First 5 participants will receive a lower dose of cord-blood derived Wharton's jelly mesenchymal stem cells (MSCTC-0010) and they will be observed for 42 days after the dose for treatment-related serious adverse events (TRSAE) and response.
  Cohort 2: Second 5 participants will receive an increased dose of MSCTC-0010 and will be observed for 42 days after the dose for TRSAE and response.
  Interventions: Biological: MSCTC-0010 Dose Escalation

INTERVENTIONS:
Biological: MSCTC-0010 Dose Escalation — Cohort 1: 2.0 × 106 cells per kilogram (cells/kg) body weight, given on day 0 and on day 7 in Participants having de novo High Risk Acute or Steroid Refractory Acute Graft Versus Host Disease (HR/SR aGvHD)
  Cohort 2: 10 × 106 cells/kg of body weight, given on day 0 and on day 7 in Participants having de novo HR/SR aGvHD
  Other Names: MSCTC-0010

SUMMARY:
This study evaluates the safety and effectiveness of two different doses of umbilical cord derived, ex-vivo cultured and expanded Wharton's jelly mesenchymal stem cells (MSCTC-0010) in the treatment of acute Graft versus Host Disease (aGVHD). The first 5 participants enrolled in the study will receive a lower dose of MSCTC-0010. If none of the first 5 participants have treatment-related serious adverse events (TRSAEs) for 42 days, then the next 5 participants will receive a slightly higher dose of MSCTC-0010.

DETAILED DESCRIPTION:
The curative potential of Allogeneic hematopoietic stem cell transplantation (allo-HCT), when applied as a therapy in the management of hematologic malignancies, specifically, derives from an immunologically driven, graft-versus-tumor effect mediated principally by donor T-cells, and is associated with a lesser risk for relapse when compared to high dose chemo-radio therapy and autologous HCT. Donor derived T-cells are also responsible for mediating the occurrence of GVHD, a common transplant-related complication, affecting a significant percentage of patients undergoing allo-HCT leading to the destruction of host tissues. The standard initial treatment for both acute and chronic GVHD is steroid-based therapy. Unfortunately, many of these patients will become resistant to steroid therapy and will subsequently be treated with second-line immunosuppressive agents. De novo high-risk aGVHD and steroid-refractory aGVHD portends a very poor prognosis; second-line agents frequently prove ineffective, and as a result, survival is < 10% at 5 years. Therefore, alternative therapies are needed to treat aGVHD following allo-HCT, particularly in the setting of de novo high-risk acute or steroid-resistant disease.

Due to the large numbers of Mesenchymal stem cells (MSC) that can be obtained from the umbilical cord, the availability of this tissue, their higher growth rates and expansion capacity, and their immune properties, including: (1) low immunogenicity and lack of stimulation of allogeneic T-lymphocyte proliferation, (2) suppression of the proliferation of activated T-lymphocytes, (3) increased production of regulatory T-cells, and (4) a shift in the immune response towards tolerance, Wharton's jelly mesenchymal stem cells (WJMSC) may be a preferred option for MSC.

The rationale for cell dosing in this protocol is based on published data from Kebriaei, et al. Dosing at 2 × 10^6 MSC/kg body weight produced a complete response in 87.5% of the treated patients. Dosing at a level 4 times higher (8 × 10^6 MSC/kg body weight) produced no improvement in complete response results. However, the higher dose produced some partial response and no patient failed to respond to therapy. Therefore, the Phase I study for MSCTC-0010 is designed to increase the dose of WJMSC from 2 × 10^6 MSC to 10 × 10^6 MSC/kg body weight, assuming no dose-limiting toxicity (DLT) is observed at the lower dose.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18 years of age and ≤ 75 years of age.
* Women of child-bearing potential and men with partners of child-bearing potential must agree to practice sexual abstinence, or to use two forms of adequate contraception (hormonal AND barrier method of birth control) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. If a woman becomes pregnant or suspects she is pregnant while participating in this study, she should inform her treating physician immediately.

  * A woman of child-bearing potential is any female (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

    * Has not undergone a hysterectomy or bilateral oophorectomy; OR
    * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)
  * Men of child-bearing potential must not donate sperm while on this study and for 90 days after their last study treatment.
  * NOTE: Acceptable forms of birth control are listed below:

    * One Barrier method (cervical cap with spermicide plus male condom; diaphragm with spermicide plus male condom) PLUS
    * Hormonal method (oral contraceptives, implants, or injections) or an intrauterine device (e.g., Copper-T).
* Participant must have de novo HR or steroid refractory, Grade II-IV aGVHD as defined in Appendix 1. NOTE: Biopsy at screening only for evaluation of aGVHD is not mandatory, but is recommended when feasible. Enrollment should not be delayed awaiting biopsy results.
* Participant must have received an allogenic transplant at Kansas University Cancer Center/University of Kansas Medical Center (KUCC / KUMC).

Exclusion Criteria:

* Participants may not have received any other investigational agent used to treat acute GVHD for 30 days prior to enrollment.
* Participant has any underlying or current medical or psychiatric condition that, in the opinion of the Investigator, would interfere with the evaluation of the participant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-07-09 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
proportion of participants who have a TRSAE after infusion of MSCTC 0010 | 45 days
  TRSAE is defined as a serious adverse event (SAE) that has a "probable" or "definite" relation to the MSCTC-0010 infusion. This study will use the descriptions and grading scales from Common Terminology Criteria for Adverse Events version 4.03 (CTCAE v4.03) for hematologic and non-hematologic toxicities.

SECONDARY OUTCOMES:
Proportion of participants who achieve a complete response (CR) of aGVHD by study day 42 | 42 days
  Complete response is defined as a complete resolution of GVHD.
Proportion of participants with improvement of GVHD in 1 or more organs involved with GVHD by day 42 | 42 days
  GVHD will be graded by organ (skin, liver, and gastrointestinal [GI])
Occurrence of addition of escalated immunosuppressive therapy by day 90 | 90 days
  Starting at the day 14 evaluation, if the acute GVHD continues to be unresponsive or worsens, additional agents or changes in immunosuppresive therapy will be at discretion of the Investigator per institutional standards.
Occurrence of Formation of ectopic tissue foci at day 90 | 90 days
  Defined as ectopic tissue formation of greater than 1.0 centimeter (cm) evaluated by comparison CT scan from screening to day 90.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph McGuirk, DO, Principal Investigator — The University of Kansas - Cancer Center
Locations (1):
- Kansas University Cancer Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No